CLINICAL TRIAL: NCT06693076
Title: Benchmarks in Acute Laparoscopic Cholecystectomy - a National Registry Study
Brief Title: Benchmarks in Acute Laparoscopic Cholecystectomy
Status: Completed | Type: Observational
Sponsor: Region Östergötland (Other)
Responsible Party: Principal Investigator, Ebba Kihlstedt Pasquier, MD, Region Östergötland
Other Study IDs: 2024-06020-02
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Gallbladder; Gall Stones (&Amp; [Calculus - Gall Bladder]); Gall Stone; Gallbladder Inflammation
Keywords: laparoscopic cholecystectomy; benchmarking; surgical outcomes; reference values; quality improvement
MeSH Terms: conditions — Gallstones; Cholecystitis | interventions — Cholecystectomy, Laparoscopic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Acute laparoscopic cholecystectomy: Patients with gallbladder inflammation. ERCP may be involved if a gallstone is detected in the common bile duct perioperatively.
  Interventions: Procedure: Laparoscopic cholecystectomy

INTERVENTIONS:
Procedure: Laparoscopic cholecystectomy — The intervention in this study is urgent, not elective. The conditions for the surgery are therefore different: any time of day, the surgeon on shift, the state of the patients.

SUMMARY:
The aim of this observational cohort study is to define peri- and postoperative reference values for acute laparoscopic cholecystectomy, using the achievable benchmarks of care methodology (ABC™). Another aim is to develop adjusted reference values for groups with a risk factor of severe postoperative complications. The goal is to spur quality improvement initiatives.

DETAILED DESCRIPTION:
The data source is the Swedish patient registry GallRiks, a prospective quality registry for gallbladder surgery and endoscopic retrograde cholangio-pancreatography (ERCP). The time frame will be 2015-2023. Register variables related to surgical quality will be analyzed, such as postoperative complications, perioperative adverse events, surgical duration and length of stay. The study will analyze data for the time of surgery and up to 30 days afterwards. As the researchers do not yet have the data available, the exact number of enrolled participants can not yet be given.

ELIGIBILITY:
Inclusion Criteria:

* adults ≥ 18 years of age
* laparoscopic acute cholecystectomy

Exclusion Criteria:

* other indications than acute cholecystitis will be excluded
* cholecystectomy due to malignancy
* other organ surgery performed at the same occasion
* previous upper gastrointestinal surgery
* single port access
* robotic surgery
* no data concerning surgical intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with gallbladder inflammation.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Benchmark values of acute laparoscopic cholecystectomy | Day of surgery
  The study will use the ABC methodology to identify reference values of surgical duration (minutes), perioperative cholangiography, conversion to open surgery and adverse events
Postoperative benchmark values of acute laparoscopic cholecystectomy | 0-30 days after surgery
  The study will use the ABC methodology to identify reference values of postoperative variables: hospital length of stay (days), abscess/infection, bleeding, biliary leakage, readmission, reoperation

SECONDARY OUTCOMES:
Adjusted benchmarks for severe complications | 0-30 days after surgery
  Univariable and multivariable logistic regression analysis will be performed to detect any risk factor for severe complications after acute laparoscopic cholecystectomy. The factors to be investigated are body mass index (kg/m2), age (years), gender, smoking, cardiovascular disease, pulmonary disease, diabetes, immunosuppressive treatment, and treatment with anticoagulants. Adjusted benchmarks will be calculated for factor(s) that in multivariable logistic regression analysis are identified as individual risk factor(s).